CLINICAL TRIAL: NCT05061550
Title: A Phase II, Open-label, Multicentre, Randomised Study of Neoadjuvant and Adjuvant Treatment in Patients With Resectable, Early-stage (II to IIIB) Non-small Cell Lung Cancer (NeoCOAST-2)
Brief Title: Neoadjuvant and Adjuvant Treatment in Resectable Non-small Cell Lung Cancer
Acronym: NeoCOAST-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9077C00001; 2023-508852-21-00 (Registry Identifier: CTIS); 2021-003369-37 (EudraCT Number)
Record Dates: First submitted 2021-09-20; First posted 2021-09-29 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Lung Cancer; early-stage; Durvalumab; Oleclumab; Monalizumab; AZD0171; Datopotamab Deruxtecan; Neoadjuvant; Adjuvant; Chemotherapy; Volrustomig; Rilvegostomig
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — durvalumab; monalizumab; Carboplatin; Cisplatin; Pemetrexed; CP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Arm 1: Oleclumab + Durvalumab + Platinum doublet chemotherapy (CTX) (Experimental): Participants will receive Durvalumab + Oleclumab + CTX as neoadjuvant treatment and Durvalumab + Oleclumab as adjuvant treatment.
  Participants will receive one of the following chemotherapy regimens, based on the tumour histology and Investigator's discretion, as part of their treatment regimen prior to surgery:
  Carboplatin/Paclitaxel Pemetrexed/Cisplatin Pemetrexed/Carboplatin
  Interventions: Drug: Durvalumab; Drug: Oleclumab; Drug: Pemetrexed/Cisplatin; Drug: Pemetrexed/Carboplatin; Drug: Carboplatin/Paclitaxel
- Arm 2: Monalizumab + Durvalumab + CTX (Experimental): Participants will receive Durvalumab + Monalizumab + CTX as neoadjuvant treatment and Durvalumab + Monalizumab as adjuvant treatment.
  Participants will receive one of the following chemotherapy regimens, based on the tumour histology and Investigator's discretion, as part of their treatment regimen prior to surgery:
  Carboplatin/Paclitaxel Pemetrexed/Cisplatin Pemetrexed/Carboplatin
  Interventions: Drug: Durvalumab; Drug: Monalizumab; Drug: Pemetrexed/Cisplatin; Drug: Pemetrexed/Carboplatin; Drug: Carboplatin/Paclitaxel
- Arm 3: Volrustomig (Dose Exploration) + CTX (Experimental): Participants will receive Volrustomig + CTX as neoadjuvant treatment and Volrustomig as adjuvant treatment.
  Participants will receive one of the following chemotherapy regimens, based on the tumour histology and Investigator's discretion, as part of their treatment regimen prior to surgery:
  Carboplatin/Paclitaxel Pemetrexed/Cisplatin Pemetrexed/Carboplatin
  Interventions: Drug: Pemetrexed/Cisplatin; Drug: Pemetrexed/Carboplatin; Drug: Carboplatin/Paclitaxel; Drug: Volrustomig
- Arm 4: Dato-DXd + durvalumab + single agent platinum (Experimental): Participants will receive Dato-DXd + durvalumab + single agent platinum as neoadjuvant treatment and durvalumab as adjuvant treatment.
  Participants will receive one of the following chemotherapy regimens, based on physician choice of as part of their treatment regimen prior to surgery:
  Carboplatin or Cisplatin
  Interventions: Drug: Durvalumab; Drug: Dato-DXd; Drug: Carboplatin; Drug: Cisplatin
- Arm 5: AZD0171 + durvalumab + CTX (Experimental): Participants will receive AZD0171 + durvalumab + CTX as neoadjuvant treatment and AZD0171 + durvalumab as adjuvant treatment.
  Participants will receive one of the following chemotherapy regimens, based on the tumour histology and Investigator's discretion, as part of their treatment regimen prior to surgery:
  Carboplatin/Paclitaxel Pemetrexed/Cisplatin Pemetrexed/Carboplatin
  Interventions: Drug: Durvalumab; Drug: AZD0171; Drug: Pemetrexed/Cisplatin; Drug: Pemetrexed/Carboplatin; Drug: Carboplatin/Paclitaxel
- Arm 6: Rilvegostomig + CTX (Experimental): Participants will receive Rilvegostomig + CTX as neoadjuvant treatment and Rilvegostomig as adjuvant treatment.
  Participants will receive one of the following chemotherapy regimens, based on the tumour histology and Investigator's discretion, as part of their treatment regimen prior to surgery:
  Carboplatin/Paclitaxel Pemetrexed/Cisplatin Pemetrexed/Carboplatin
  Interventions: Drug: Pemetrexed/Cisplatin; Drug: Pemetrexed/Carboplatin; Drug: Carboplatin/Paclitaxel; Drug: Rilvegostomig
- Arm 7: Dato-DXd + Rilvegostomig + single agent platinum (Experimental): Participants will receive Dato-DXd + Rilvegostomig + single agent platinum as neoadjuvant treatment and Rilvegostomig as adjuvant treatment.
  Participants will receive one of the following chemotherapy regimens, based on physician choice of as part of their treatment regimen prior to surgery:
  Carboplatin or Cisplatin
  Interventions: Drug: Dato-DXd; Drug: Carboplatin; Drug: Cisplatin; Drug: Rilvegostomig

INTERVENTIONS:
Drug: Durvalumab — Participants will receive Durvalumab via intravenous route.
  Other Names: MEDI4736, IMFINZI
  Arms: Arm 1: Oleclumab + Durvalumab + Platinum doublet chemotherapy (CTX); Arm 2: Monalizumab + Durvalumab + CTX; Arm 4: Dato-DXd + durvalumab + single agent platinum; Arm 5: AZD0171 + durvalumab + CTX
Drug: Oleclumab — Participants will receive Oleclumab via intravenous route.
  Other Names: MEDI9447
  Arms: Arm 1: Oleclumab + Durvalumab + Platinum doublet chemotherapy (CTX)
Drug: Monalizumab — Participants will receive Monalizumab via intravenous route.
  Other Names: IPH2201
  Arms: Arm 2: Monalizumab + Durvalumab + CTX
Drug: Dato-DXd — Participants will receive datopotamab deruxtecan (Dato-DXd) via intravenous route.
  Arms: Arm 4: Dato-DXd + durvalumab + single agent platinum; Arm 7: Dato-DXd + Rilvegostomig + single agent platinum
Drug: AZD0171 — Participants will receive AZD0171 via intravenous route.
  Arms: Arm 5: AZD0171 + durvalumab + CTX
Drug: Carboplatin — Carboplatin as chemotherapy
  Arms: Arm 4: Dato-DXd + durvalumab + single agent platinum; Arm 7: Dato-DXd + Rilvegostomig + single agent platinum
Drug: Cisplatin — Cisplatin as chemotherapy
  Arms: Arm 4: Dato-DXd + durvalumab + single agent platinum; Arm 7: Dato-DXd + Rilvegostomig + single agent platinum
Drug: Pemetrexed/Cisplatin — Pemetrexed/Cisplatin as chemotherapy
  Arms: Arm 1: Oleclumab + Durvalumab + Platinum doublet chemotherapy (CTX); Arm 2: Monalizumab + Durvalumab + CTX; Arm 3: Volrustomig (Dose Exploration) + CTX; Arm 5: AZD0171 + durvalumab + CTX; Arm 6: Rilvegostomig + CTX
Drug: Pemetrexed/Carboplatin — Pemetrexed/Carboplatin as chemotherapy
  Arms: Arm 1: Oleclumab + Durvalumab + Platinum doublet chemotherapy (CTX); Arm 2: Monalizumab + Durvalumab + CTX; Arm 3: Volrustomig (Dose Exploration) + CTX; Arm 5: AZD0171 + durvalumab + CTX; Arm 6: Rilvegostomig + CTX
Drug: Carboplatin/Paclitaxel — Carboplatin/Paclitaxel, as chemotherapy
  Arms: Arm 1: Oleclumab + Durvalumab + Platinum doublet chemotherapy (CTX); Arm 2: Monalizumab + Durvalumab + CTX; Arm 3: Volrustomig (Dose Exploration) + CTX; Arm 5: AZD0171 + durvalumab + CTX; Arm 6: Rilvegostomig + CTX
Drug: Volrustomig — Participants will receive Volrustomig via intravenous route.
  Other Names: MEDI5752
  Arms: Arm 3: Volrustomig (Dose Exploration) + CTX
Drug: Rilvegostomig — Participants will receive Rilvegostomig via intravenous route.
  Arms: Arm 6: Rilvegostomig + CTX; Arm 7: Dato-DXd + Rilvegostomig + single agent platinum

SUMMARY:
The study is intended to assess the safety and efficacy of perioperative treatment with Durvalumab in combination with Oleclumab, Monalizumab, or AZD0171 and platinum doublet chemotherapy (CTX); or Volrustomig or Rilvegostomig in combination with CTX; or Datopotamab deruxtecan (Dato-DXd) in combination with Durvalumab or Rilvegostomig and single agent platinum chemotherapy in participants with resectable, early-stage non-small cell lung cancer.

DETAILED DESCRIPTION:
This is an open-label, multi-arms, multicentre, randomised study, eligible participants will be enrolled and randomised to one of the following treatment regimens.

Arm 1: Participants will receive Oleclumab + durvalumab + CTX as neoadjuvant treatment and Oleclumab + durvalumab as adjuvant treatment.

Arm 2: Participants will receive Monalizumab + durvalumab + CTX as neoadjuvant treatment and Monalizumab + durvalumab as adjuvant treatment.

Arm 3: Participants will receive Volrustomig (Dose Exploration) + CTX as neoadjuvant treatment and Volrustomig as adjuvant treatment.

Arm 4: Participants will receive Dato-DXd + durvalumab + single agent platinum chemotherapy as neoadjuvant treatment and durvalumab as adjuvant treatment.

Arm 5: Participants will receive AZD0171 + durvalumab + CTX as neoadjuvant treatment and AZD0171 + durvalumab as adjuvant treatment.

Arm 6: Participants will receive Rilvegostomig + CTX as neoadjuvant treatment and Rilvegostomig as adjuvant treatment.

Arm 7: Participants will receive Dato-DXd + Rilvegostomig + single agent platinum chemotherapy as neoadjuvant treatment and Rilvegostomig as adjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed NSCLC patients with resectable disease (Stage IIA to Stage IIIB).
* WHO or Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ and bone marrow function.
* Provision of tumour samples (newly acquired or archival tumour tissue [≤ 6 months old]) to confirm Programmed death-ligand 1 (PD-L1) status, epidermal growth factor receptor (EGFR), or anaplastic lymphoma kinase (ALK) status.
* Adequate pulmonary function.

Exclusion Criteria:

* Participants with sensitising EGFR mutations or ALK translocations.
* Participants with baseline PD-L1 expression status <1% (Arms 6 and 7 only).
* Active or prior documented autoimmune or inflammatory disorders.
* Uncontrolled intercurrent illness, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, active bleeding diseases, serious chronic gastrointestinal conditions associated with diarrhoea, or psychiatric illness/social situations that would limit compliance with study requirement.
* History of another primary malignancy.
* Participants with small-cell lung cancer or mixed small-cell lung cancer.
* History of active primary immunodeficiency.
* History of non-infectious interstitial lung disease (ILD) ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or has suspected ILD/pneumonitis that cannot be ruled out by imaging at screening.
* Participants who have preoperative radiotherapy treatment as part of their care plan.
* Participants who require or may require pneumonectomy, segmentectomies, or wedge resections, as assessed by their surgeon at baseline, to obtain potentially curative resection of primary tumour.
* QTcF (QT interval corrected by Fridericia's formula) interval ≥ 470 ms.
* Any medical contraindication to treatment with chemotherapy as listed in the local labelling.
* Participants with moderate or severe cardiovascular disease.
* Any concurrent chemotherapy, investigational product, biologic, or hormonal therapy for cancer treatment.
* Receipt of live attenuated vaccine within 30 days prior to the first dose of study interventions.
* Prior exposure to approved or investigational immune-mediated therapy including, but not limited to, other anti-CTLA-4, anti-TIGIT (T cell immunoreceptor with Ig and ITIM domains), anti-PD-1, anti-PD-L1, and anti-PD-L2 antibodies. Participants who received agents targeting the adenosine pathway, anti-NKG2A, anti-HLA-E agents, and anti-LIF agents are also excluded. Participants who have received previous treatment with a TROP2 targeting ADC or with another ADC containing a chemotherapy agent that inhibits TOP1 activity are also excluded.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of study interventions.
* Active or uncontrolled infections including HBA, HBV, HCV, and HIV.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2030-05-09 (Estimated); Study Completion 2030-05-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with pathological complete response (pCR) | From randomization to approximately 15 weeks after the first dose of study interventions
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Until Day 90 after the last dose of study interventions (Up to approximately 3 years)

SECONDARY OUTCOMES:
Number of participants experiencing an event-free survival (EFS) event | Up to approximately 3 years
Number of participants experiencing a disease-free survival (DFS) event | Up to approximately 3 years
Number of participants having surgical resection | From randomization to approximately 15 weeks after the first dose of study interventions
Number of participants with major pathological response (mPR) | From randomization to approximately 15 weeks after the first dose of study interventions
Number of participants with Objective response rate (ORR) | From randomization to approximately 15 weeks after the first dose of study interventions
Overall survival (OS) | Up to approximately 3 years
Serum concentration of study interventions (Durvalumab/Oleclumab/Monalizumab/Volrustomig/Rilvegostomig) | From randomization to last dose of study interventions (Up to approximately 3 Years)
Number of participants with anti-study drug antibodies (ADA) | From randomization to 3 months after last dose of study interventions (Up to approximately 3 Years)
Baseline PD-L1 expression | At Screening/ baseline
Changes in circulating tumour DNA (ctDNA) | From randomization to up to 24 months after last dose of study interventions (Up to approximately 3 Years)

CONTACTS AND LOCATIONS:
Overall Officials: Tina Cascone, MD, Principal Investigator — MD Anderson Cancer Center Houston, TX 77030
Locations (80):
- United States (21):
  - Research Site, Little Rock, Arkansas
  - Research Site, Los Angeles, California
  - Research Site, Oakland, California
  - Research Site, New Haven, Connecticut
  - Research Site, Stuart, Florida
  - Research Site, Gainesville, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Saint Louis Park, Minnesota
  - Research Site, Omaha, Nebraska
  - Research Site, Buffalo, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Chattanooga, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, Edmonds, Washington
  - Research Site, Seattle, Washington
- Belgium (4):
  - Research Site, Charleroi
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Roeselare
- Canada (3):
  - Research Site, Edmonton, Alberta
  - Research Site, Winnipeg, Manitoba
  - Research Site, Montreal, Quebec
- France (8):
  - Research Site, Avignon
  - Research Site, Bobigny
  - Research Site, Bordeaux
  - Research Site, Limoges
  - Research Site, Rennes
  - Research Site, Rouen
  - Research Site, Suresnes
  - Research Site, Toulon
- Hungary (4):
  - Research Site, Kecskemét
  - Research Site, Székesfehérvár
  - Research Site, Tatabánya
  - Research Site, Törökbálint
- Ireland (2):
  - Research Site, Dublin
  - Research Site, Galway
- Italy (13):
  - Research Site, Aviano
  - Research Site, Brescia
  - Research Site, Catanzaro
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Monza
  - Research Site, Padua
  - Research Site, Perugia
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Rozzano
- Portugal (2):
  - Research Site, Lisbon
  - Research Site, Porto
- South Korea (5):
  - Research Site, Busan
  - Research Site, Chungcheongbuk-do
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (11):
  - Research Site, A Coruña
  - Research Site, Alicante
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Málaga
  - Research Site, Reus
  - Research Site, Seville
  - Research Site, Terrassa
  - Research Site, Valencia
- Taiwan (4):
  - Research Site, Liuying
  - Research Site, New Taipei City
  - Research Site, Tainan
  - Research Site, Taipei
- Turkey (Türkiye) (3):
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- [Derived] Cascone T, Bonanno L, Guisier F, Insa A, Liberman M, Bylicki O, Livi L, Egenod T, Corre R, Kim DW, Garcia Campelo MR, Provencio Pulla M, Shim BY, Metro G, Bennouna J, Bielska AA, Yohannes AR, He Y, Dowson A, Kar G, McGrath L, Kumar R, Grenga I, Spicer J, Forde PM. Perioperative durvalumab plus chemotherapy plus new agents for resectable non-small-cell lung cancer: the platform phase 2 NeoCOAST-2 trial. Nat Med. 2025 Aug;31(8):2788-2796. doi: 10.1038/s41591-025-03746-z. Epub 2025 May 31. PMID 40450142
- See also: Lung Cancer Study Locator details (for US) — https://www.lungcancerstudylocator.com/trial/listing/305617